CLINICAL TRIAL: NCT00111553
Title: Randomized, Double-Blind, Adjuvant- and Placebo-Controlled, Dose-Escalating Study to Evaluate Safety, Tolerability, and Immunogenicity of Leish-111f + MPL-SE Vaccine With Meglumine Antimoniate (Glucantime) in Cutaneous Leishmaniasis
Brief Title: Study to Evaluate the Leish-111F + MPL-SE Vaccine in the Treatment of Cutaneous Leishmaniasis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Access to Advanced Health Institute (AAHI) (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IDRI-LCVTC-101
Record Dates: First submitted 2005-05-23; First posted 2005-05-24 (Estimated); Last update posted 2007-02-15 (Estimated); Status verified 2007-02

CONDITIONS: Leishmaniasis, Cutaneous
Keywords: Leishmaniasis; Subunit vaccine; Therapeutic; T cell; Antimony
MeSH Terms: conditions — Leishmaniasis, Cutaneous; Leishmaniasis

INTERVENTIONS:
Biological: Leish-111f + MPL-SE vaccine

SUMMARY:
This study will evaluate the safety of the Leish-111f + MPL-SE vaccine in adult patients with cutaneous leishmaniasis.

DETAILED DESCRIPTION:
Cutaneous leishmaniasis is a disfiguring infection that can progress to mucosal leishmaniasis, a more serious and possibly fatal form of leishmania infection. All available medical therapies require weeks of treatment and cause significant toxicity. In Brazil, a standard therapy is Glucantime treatment, administered in cycles of 10 consecutive, once daily, intramuscular injections (Glucantime 10 mg/kg, maximum of 850 mg), followed by 11 consecutive days without Glucantime injections (rest days). At the completion of each cycle, a study physician examines the patient to determine if a further cycle of Glucantime treatment is indicated.

It appears that Leishmania infections can be eliminated by T helper 1 immune responses. This finding argues that a vaccine that augments cutaneous leishmaniasis patients' T helper 1 response will eliminate the infection and disease. This study is a phase 1, randomized, double-blind, placebo controlled, sequential dose-escalating trial to evaluate the safety and immunogenicity of three injections of 5, 10, or 20 μg of Leish-111f protein + 25 μg of MPL-SE adjuvant given at 4 week intervals as an adjunct to the standard chemotherapy with Glucantime cycles, as described above in patients with cutaneous leishmaniasis.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of cutaneous leishmaniasis defined as positive identification of parasite from lesion biopsy
* Normal lab values and electrocardiogram (ECG)
* Negative for HIV, hepatitis B and C, and Chagas disease

Exclusion Criteria:

* Nine or more active cutaneous lesions
* Lesion diameter >60mm
* Previous exposure to Leishmania vaccines or to MPL-SE
* Pregnant or breastfeeding female

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45
Dates: Start 2004-10; Study Completion 2006-08

PRIMARY OUTCOMES:
Occurrence of dose limiting toxicity
Adverse events

SECONDARY OUTCOMES:
IgG and T-cell response to Leish-111f vaccine
Leish-111f skin test reactivity
Safety of the vaccine with respect to the clinical course of cutaneous leishmaniasis

CONTACTS AND LOCATIONS:
Overall Officials: Evaldo Nascimento, MD, Principal Investigator — Federal University of Minas Gerais; Franco M Piazza, MD, MPH, Study Director — Infectious Disease Research Institute (IDRI)
Locations (2):
- Brazil (2):
  - Universidade Federal de Minas Gerais, Belo Horizonte, Minas Gerais
  - Ambulatório de Leishmanioses da Secretaria Municipal da Saude de Januária, Januária, Minas Gerais